CLINICAL TRIAL: NCT00003797
Title: Herceptin (NSC #688097) and Gemcitabine for Metastatic Pancreatic Cancers That Overexpress HER-2/NEU
Brief Title: Gemcitabine and Monoclonal Antibody Therapy in Treating Patients With Metastatic Cancer of the Pancreas
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Brown University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000066940; BRUOG-PA-77; NCI-T98-0067
Record Dates: First submitted 1999-11-01; First posted 2003-05-02 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2002-12

CONDITIONS: Pancreatic Cancer
Keywords: recurrent pancreatic cancer; stage IV pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Trastuzumab; Gemcitabine

INTERVENTIONS:
Biological: trastuzumab
Drug: gemcitabine hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Monoclonal antibodies such as trastuzumab can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells. Combining monoclonal antibody therapy with chemotherapy may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of gemcitabine and trastuzumab in treating patients who have metastatic cancer of the pancreas that overexpresses HER2/neu.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the response rate and survival of patients with metastatic pancreatic cancer and overexpression of HER2/neu treated with gemcitabine and trastuzumab.
* Determine the toxic effects of this regimen in these patients.

OUTLINE: This is a multicenter study.

Patients receive gemcitabine IV over 30 minutes once weekly during weeks 1-7. Patients receive trastuzumab IV over 90 minutes once during week 1 and trastuzumab IV over 30-90 minutes once weekly during weeks 2-8.

Patients with stable or responding disease receive gemcitabine IV over 30 minutes once weekly during weeks 1-3 and trastuzumab IV over 30 minutes once weekly during weeks 1-4. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months for 1 year and then every 6 months thereafter.

PROJECTED ACCRUAL: A maximum of 41 patients will be accrued for this study over 18-24 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven metastatic pancreatic cancer with overexpression of HER2/neu
* Patients in whom there is inadequate tissue to evaluate for HER2/neu overexpression but who have elevated serum HER2/neu antigen levels are eligible
* Radiographically measurable disease

  * May have metastatic disease in which primary lesion is measurable but metastatic lesions are not measurable
  * Ascites is not measurable

PATIENT CHARACTERISTICS:

Age:

* Over 18

Performance status:

* ECOG 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Granulocyte count at least 1,500/mm3
* Platelet count at least 100,000/mm3

Hepatic:

* Bilirubin no greater than 3.0 mg/dL

  * Greater than 3 times normal if increase in bilirubin is due to biliary obstruction from tumor as long as biliary system is stented or bypassed and bilirubin, SGOT, or SGPT is stable or decreasing
* SGOT no greater than 3 times normal

  * No greater than 5 times normal if liver metastases present OR
  * Greater than 5 times normal if increase in SGOT or SGPT is due to biliary obstruction from tumor as long as biliary system is stented or bypassed and biliary SGOT or SGPT is stable or decreasing

Renal:

* Creatinine no greater than 2.0 mg/dL

Cardiovascular:

* No unstable angina
* No prior congestive heart failure
* No prior myocardial infarction
* LVEF at least 45% by MUGA or echocardiogram

Other:

* Not pregnant
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior trastuzumab
* No concurrent growth factors

Chemotherapy:

* No prior anthracyclines
* No prior gemcitabine except prior low dose (no greater than 300 mg/m2/week) gemcitabine with radiotherapy
* At least 6 months since prior adjuvant therapy
* More than 2 weeks since other prior chemotherapy
* No other concurrent cytotoxic chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* See Chemotherapy
* More than 2 weeks since prior radiotherapy
* No concurrent radiotherapy

Surgery:

* Not specified

Other:

* No other concurrent investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Estimated)
Dates: Start 1999-03

CONTACTS AND LOCATIONS:
Overall Officials: Howard Safran, MD, Study Chair — Brown University
Locations (12):
- United States (12):
  - Rush-Presbyterian-St. Luke's Medical Center, Chicago, Illinois
  - New England Medical Center Hospital, Boston, Massachusetts
  - St. Elizabeth's Medical Center, Boston, Massachusetts
  - Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Mount Sinai Medical Center, NY, New York, New York
  - University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - Memorial Hospital of Rhode Island, Pawtucket, Rhode Island
  - Rhode Island Hospital, Providence, Rhode Island
  - Roger Williams Medical Center/BUSM, Providence, Rhode Island
  - Brown University Oncology Group, Providence, Rhode Island
  - University of Texas - MD Anderson Cancer Center, Houston, Texas